CLINICAL TRIAL: NCT04370184
Title: Ultrasound Imaging of the Brachial Plexus Sheath and Its Fascial Compartments at the Costoclavicular Space and Infraclavicular Fossa
Brief Title: USG Imaging of Brachial Plexus Sheath & Its Fascial Compartments at Costoclavicular Space & Infraclavicular Fossa
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof Manoj K Karmakar, Professor, Chinese University of Hong Kong
Other Study IDs: HD BPS Protocol Version 1
Record Dates: First submitted 2020-04-29; First posted 2020-04-30 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Musculoskeletal Diseases or Conditions
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Ultrasound guided Costoclavicular Brachial Plexus Block — Ultrasound images from patients scheduled for upper limb surgery under costoclavicular brachial plexus block (one kind of regional anesthesia) have been routinely collected at our institute. These images will be reviewed.

SUMMARY:
The existence of the brachial plexus sheath (BPS) and its septae and compartments has been a subject of debate and controversy. Numerous cadaver studies indicate that BPS is present while other researchers based on limited clinical data suggest none. Nevertheless, cumulative evidence over the last six decades indicate that it is multi-layered, fibrous and a web-like connective tissue that is derived from the deep cervical fascia and fused with the deep fascia of the arm The BPS completely envelopes that neurovascular bundle and filed with loose connective tissue and fat. It is a multi-compartment structure in the axilla with each nerve having a separate compartment, that communicate with each other. Some studies suggested that the septae affect the spread of local anesthetic during an axillary or infraclavicular brachial plexus block, while some suggest the opposite. With the use of ultrasound imaging, researchers found the presence of this connective tissue septum within the BPS at the costoclavicular space and infraclavicular fossa. The septum is visualized as a linear hyperechoic band on ultrasound imaging and when present appears to reduce the spread of the drugs during brachial plexus block. Yet the anatomy is poorly seen with the previous generation of ultrasound imaging. The aim of this study is to define the connective tissue (fascial) layers that surround the brachial plexus and its septum at the infraclavicular fossa by reviewing our archived high definition ultrasound images of 100 patients who had successfully undergone the ultrasound guided brachial plexus block over a 5 year period (2013 to 2018).

DETAILED DESCRIPTION:
This is a retrospective study reviewing archived high definition ultrasound images as multiple short video loops (6 seconds) in avi format from 100 adult patients who had undergone ultrasound guided costoclavicular brachial plexus block for surgical anesthesia for their upper limb surgery over a 5 year period, from April 2013 to April 2018 by three experienced anesthesiologists. Demographics data such as age, gender, body mass index, ASA Physical Classification System, local anesthetic drug used and mode of anesthesia can be retrieved from patients' record or Clinical Management System. No direct contact nor intervention will be done to the patients in this study, so waiver of patient informed consent has been sought. There will be no patients' data in any of the ultrasound images as the ultrasound video loops for the costoclavicular brachial plexus block are routinely saved anonymously for all patients. All information related to the patients will be kept confidential and they will not be identified in any form in future publications.

ELIGIBILITY:
Inclusion Criteria:

* Archived high definition ultrasound images (datasets) as multiple short video loop (6 seconds) in avi format from 100 adult patients who had undergone ultrasound guided costoclavicular brachial plexus block for surgical anesthesia during forearm or hand surgery, over a 5 year period, from April 2013 to April 2018 will be retrieved for review.

Exclusion Criteria:

* > 70 years old, BMI >30, ASA physical status > III, and with previous history surgery over the infraclavicular fossa

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 adult patients who had undergone ultrasound guided costoclavicular brachial plexus block for surgical anesthesia during forearm or hand surgery over a 5 year period, from April 2013 to April 2018.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
ultrasound visibility of the anatomical structures around the neck | 1 day (will be reviewed once)
  Positive or negative ultrasound visibility (yes or no response) of a given anatomical structure (pectoralis major muscle, subclavius muscle, serratus anterior muscle, costoclavicular space, axillary artery, lateral, medial and posterior cords of the brachial plexus, brachial plexus space (BPS), septum within the BPS, and the anterior & posterior compartment) will be agreed upon by consensus among the three outcome assessors. If a structure is visible the quality of ultrasound visibility will be assessed using a 4-point Likert scale (0=not visible, 1=hardly visible, 2=well visible, 3=very well visible). The total ultrasound visibility score (UVS, maximum score possible is 36 at the costoclavicular space and 33 at the lateral infraclavicular fossa will thereby computed.

CONTACTS AND LOCATIONS:
Overall Officials: Manoj K Karmakar, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hosptial, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Areeruk P, Karmakar MK, Reina MA, Mok LYH, Sivakumar RK, Sala-Blanch X. High-definition ultrasound imaging defines the paraneural sheath and fascial compartments surrounding the cords of the brachial plexus at the costoclavicular space and lateral infraclavicular fossa. Reg Anesth Pain Med. 2021 Jun;46(6):500-506. doi: 10.1136/rapm-2020-102304. Epub 2021 Apr 2. PMID 33811182